CLINICAL TRIAL: NCT06718764
Title: Evaluating the Feasibility of Utilizing a Novel Brain Activity Monitor in the Neurosciences Intensive Care Unit
Brief Title: Neurosteer Bedside Monitoring System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Neurosteer Ltd. (Industry)
Responsible Party: Principal Investigator, Neha Dangayach, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY-23-00018
Record Dates: First submitted 2024-07-15; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Delirium; Sedation; Agitation
MeSH Terms: conditions — Delirium; Psychomotor Agitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- NSICU Patients with Acute Neurological Injuries (ANI) (Active Comparator): ANI are participants having Acute Ischemic Stroke (AIS), Intracerebral Hemorrhage, Subarachnoid Hemorrhage (SAH), Status Epileptics, Traumatic Brain Injury (TBI), Brain Tumors, Meningitis/encephalitis, post cardiac arrest hypoxic ischemic encephalopathy. All participants will be set up with the Neurosteer bedside monitoring system.
  Interventions: Device: Neurosteer's single-channel EEG monitoring device
- NSICU Patients without Acute Neurological Injuries (ANI) (Active Comparator): Participants without ANI to have neuromuscular disorders such as myasthenia gravis, spine surgery, septic shock, acute respiratory distress syndrome, and Hemorrhagic shock ex. from gastrointestinal bleeding. All participants will be set up with the Neurosteer bedside monitoring system.
  Interventions: Device: Neurosteer's single-channel EEG monitoring device

INTERVENTIONS:
Device: Neurosteer's single-channel EEG monitoring device — Neurosteer device will be attached to participants forehead and readings will be collected for the duration of their NSICU stay.
  Neurosteer auditory stimulation will be done 3-4 times a day to coincide with RASS and 1-2 times a day to coincide with CAM-ICU. The research team will correlate collected hourly RASS and CAM-ICU assessments with Neurosteer derived signals and parameters.

SUMMARY:
The purpose of this study is to evaluate the clinical utility of Neurosteer's brain monitoring platform for monitoring delirium, sedation, and agitation in intubated and sedated ICU patients. The research team will be conducting a single-site study. The research team will enroll 100 patients admitted to the NSICU. 50 of these patients will have Acute Neurological Injuries (ANI) and the other 50 will not have an ANI. All enrolled patients will receive the intervention, the Neurosteer brain monitoring device.

The study intervention consists of the use of Neurosteer's innovative single-channel EEG monitoring device to determine if there is a good correlation and agreement between their signals/parameters to RASS, CAM-ICU, and continuous EEG monitoring readings. The Neurosteer device will be attached to their forehead and readings will be collected for the duration of their NSICU stay. The research team will adapt the current physical methods of detecting the depth of anesthesia i.e. through the Richmond Agitation-Sedation Scale (RASS) & CAM-ICU, to auditory stimulation, which will be delivered through earphones with no physical contact, with the aim of achieving a high correlation between the methods. RASS and CAM-ICU will be collected hourly as standard of care and Neurosteer auditory stimulation will be done 3-4 times a day to coincide with RASS and 1-2 times a day to coincide with CAM-ICU. The research team will correlate collected hourly RASS and CAM-ICU assessments with Neurosteer derived signals and parameters.

DETAILED DESCRIPTION:
In the study population of sedated, intubated critically ill patients, the research team hypothesize the following:

* Neurosteer's derived signals and parameters will be correlated to and will have at least fair agreement with the Richmond Agitation Sedation Scale (RASS) for measuring depth of sedation.
* Neurosteer's derived signals and parameters will be correlated to and have at least fair agreement with the Confusion Assessment Method (CAM-ICU) to screen for and diagnose delirium.
* For enrolled patients undergoing cEEG monitoring as standard of care, the detection of burst suppression, seizures, and ictal-interictal continuum between Neurosteer's derived signals and parameters and continuous EEG monitoring readings will be correlated and have at least fair agreement.
* There will be no significant difference in the correlations determined in our primary objective between NSICU patients with and without ANI.

The research team will be conducting a single-site study to evaluate these hypotheses. The research team will enroll 100 patients admitted to the NSICU. 50 of these patients will have an ANI and the other 50 will not have an ANI. The research team will define ANI as subjects having Acute Ischemic Stroke (AIS), Intracerebral Hemorrhage, Subarachnoid Hemorrhage (SAH), Status Epileptics, Traumatic Brain Injury (TBI), Brain Tumors, Meningitis/encephalitis, post cardiac arrest hypoxic ischemic encephalopathy. The research team will define subject without ANI to have neuromuscular disorders such as myasthenia gravis, spine surgery, septic shock, acute respiratory distress syndrome, and Hemorrhagic shock ex. from gastrointestinal bleeding. The research team will obtain written informed consent from all patients and/or their Legally Authorized Representative (LAR) to conduct the study. All enrolled patients will receive the intervention, the Neurosteer brain monitoring platform. Intra-individual comparisons will be made between standard of care assessments and the findings of the Neurosteer device. Inter-individual comparisons between patients with and without ANI will also be made. Statistical analyses will be conducted halfway through study enrollment and upon completion of enrollment and data entry. The study intervention will span the duration of the patient's admission in the NSICU. Patients will be screened for consented and screened for eligibility as they get admitted to the NSICU.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form from patient and/or LAR, including stated willingness to comply with all study procedures and availability for the duration of the study
* Any assigned sex at birth, including individuals who are transgender or intersex
* Age 18 years or older
* Mechanically ventilated patients with an anticipated LOS >/=48 hours on any sedative drips including propofol, midazolam, dexmedetomidine, fentanyl, dialudid, ketamine

Exclusion Criteria:

* Has known hearing problems and usage of hearing aids
* Has a rash on forehead
* History of polysubstance abuse
* Severe dementia
* Anticipated Withdrawing Life-Sustaining Therapy (WLST) within the next 24-48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Sedation as measured by Richmond Agitation Sedation Scale | 3-4 times daily throughout participants NSICU stay (average 14 days)
  Richmond Agitation Sedation Scale (RASS) for measuring the depth of sedation in sedated, intubated critically ill patients. RASS scoring -5 to +4, is a valid and reliable instrument to assess level of sedation and agitated behavior during sedation, where higher scores indicate higher levels of agitation.
  4 Combative, violent, danger to staff 3 Pulls or removes tube(s) or catheters; aggressive 2 Frequent non-purposeful movement
  1 Anxious, apprehensive, but not aggressive 0 Alert and calm
  1. Awakens to voice (eye opening/contact) >10 sec
  2. Light sedation, briefly awakens to voice (eye opening/contact) <10 sec
  3. Moderate sedation, movement or eye opening. No eye contact
  4. Deep sedation, no response to voice, but movement or eye opening to physical stimulation
  5. Unarousable, no response to voice or physical stimulation

SECONDARY OUTCOMES:
Delirium as measured by Confusion Assessment Method (CAM) | 1-2 times daily throughout participants NSICU stay (average 14 days)
  Confusion Assessment Method (CAM) for screening and diagnosing delirium in intubated, sedated critically ill patients. The CAM consists of 4 features: 1-Onset, 2-Inattention, 3-Disorganized thinking, and 4-altered level of consciousness. The diagnosis of delirium by CAM is based on the presence of features 1 and 2, and either 3 or 4.

CONTACTS AND LOCATIONS:
Overall Officials: Neha S Dangayach, MD, MSCR, FNCS, FAAN, DCE'21, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
The research team will only share aggregated, de-identified data with the sponsor solely for the purpose of analyzing correlations.